CLINICAL TRIAL: NCT07393984
Title: Effect of Digital Self-Monitoring on Patient Engagement and Clinical Outcomes in Severe Asthma: A Randomized Controlled Pilot Study
Brief Title: Digital Self-Monitoring in Severe Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Pharmacy "Victor Babes" Timisoara (Other)
Responsible Party: Principal Investigator, Norbert Wellmann, MD, Pulmonology Resident, PhD Student, University of Medicine and Pharmacy "Victor Babes" Timisoara
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AIOCARE-SEV-ASTHMA
Record Dates: First submitted 2026-01-25; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Severe Asthma; Asthma
Keywords: Severe asthma; Telemedicine; Digital health; Home spirometry; Adherence; Patient engagement; Reminders; eHealth
MeSH Terms: conditions — Asthma; Patient Participation

STUDY DESIGN:
Intervention Model Description: This was a single-center, randomized, parallel-group pilot study. Participants were randomized in a 1:1 ratio to either an intervention group receiving weekly reminder messages via SMS or via the AioCare platform, or to a control group receiving standard telemedicine-based home monitoring without reminders.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Reminder) (Experimental): Adults with severe asthma who used the AioCare digital respiratory system for home spirometry and received weekly reminder messages via SMS or in-app notifications to support adherence.
  Interventions: Device: AioCare home spirometry system
- Control group (Active Comparator): Adults with severe asthma who used the AioCare digital respiratory system for home spirometry without receiving reminder messages (standard remote monitoring).
  Interventions: Device: AioCare home spirometry system

INTERVENTIONS:
Device: AioCare home spirometry system — The AioCare digital respiratory system was used to perform weekly home spirometry and to transmit lung function data to a secure telemedicine platform for remote monitoring by the study team.

SUMMARY:
This randomized controlled pilot study aimed to assess adherence to telemedicine-based home monitoring using the AioCare digital respiratory system in adults with severe asthma over a three-month period and to determine whether weekly reminder messages sent via SMS or through the AioCare platform enhanced adherence compared with standard remote monitoring.

The study was conducted at a single center in Timișoara, Romania, between October 2024 and October 2025. Thirty adult patients with severe asthma were randomized 1:1 to either an intervention group receiving weekly reminders via SMS or in-app notifications, or a control group without reminders. All participants performed weekly home spirometry for 12 weeks using the AioCare system.

The primary objective of the study was to assess adherence to telemedicine-based home monitoring over the three-month period and to evaluate the effect of weekly reminder messages on adherence compared with standard remote monitoring.

The study found that patients who received reminder messages demonstrated higher adherence to home monitoring compared with those who did not receive reminders. No device-related adverse events were reported.

DETAILED DESCRIPTION:
This study investigated telemedicine-based home monitoring in adults with severe asthma using the AioCare digital respiratory system in a real-world clinical setting.

Participants were equipped with a portable AioCare spirometry device and trained to use the associated mobile application for home measurements. The system enabled wireless transmission of spirometric data to a secure cloud-based platform, allowing remote review of patient-generated data by the study team.

After enrollment and training, patients performed regular home spirometry over a three-month monitoring period. Measurements were conducted in the patients' home environment and automatically uploaded through the AioCare platform. Data quality was assessed according to international acceptability and repeatability criteria.

One study group additionally received automated weekly reminder messages delivered via SMS or through the AioCare application, depending on technical availability and patient preference. These reminders were standardized and intended to support regular performance of home measurements. The comparator group used the same monitoring system without reminders.

Throughout the study, participants continued their usual standard-of-care treatment. No experimental medications or therapeutic interventions were introduced. Study procedures focused on remote data collection, monitoring feasibility, and patient interaction with the digital health system.

At the end of the monitoring period, patient-reported questionnaires were administered to document user experience with the telemonitoring system. Safety was monitored throughout the study, with specific attention to device-related adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of severe asthma according to GINA guidelines.
* Age ≥ 18 years.
* Ability to correctly perform spirometry maneuvers according to ATS/ERS standards after training.
* Access to a smartphone compatible with the AioCare application.
* Willingness to participate in weekly home-based spirometry monitoring and telemonitoring for three months.
* Stable maintenance asthma therapy for at least four weeks prior to enrollment.
* Ability and willingness to provide written informed consent.

Exclusion Criteria:

* Age < 18 years.
* Diagnosis of other significant respiratory diseases (including chronic obstructive pulmonary disease, interstitial lung disease, or bronchiectasis).
* Asthma exacerbation requiring hospitalization or systemic corticosteroids within the four weeks prior to enrollment.
* Severe psychiatric or cognitive impairment that could interfere with adherence to the monitoring protocol or ability to use the device independently.
* Inability to perform acceptable spirometry maneuvers despite training.
* Lack of smartphone or internet access required for AioCare telemonitoring.
* Pregnancy or breastfeeding.
* Refusal or inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Adherence to telemedicine-based home monitoring | 12 weeks
  Proportion of prescribed weekly home spirometry sessions successfully completed and transmitted via the AioCare system during the 12-week monitoring period.
Asthma control assessed by ACT | Baseline and 12 weeks
  Change in Asthma Control Test (ACT) score from baseline to week 12. The ACT is a validated 5-item questionnaire, with scores ranging from 5 to 25, where higher scores indicate better asthma control. Scores ≥20 indicate well-controlled asthma, 16-19 partially controlled, and ≤15 poorly controlled. A change of ≥3 points is considered clinically meaningful.

OTHER OUTCOMES:
Patient-reported satisfaction and engagement with the telemonitoring system | 12 weeks
  Patient-reported satisfaction and engagement will be assessed at the end of the 12-week study period using an adapted version of the mHealth App Usability Questionnaire (MAUQ). The instrument includes 10 dichotomous (Yes/No) items. Responses are coded as Yes = 1 and No = 0 and summed to generate a total score ranging from 0 to 10. Higher scores indicate greater satisfaction, perceived usefulness, and engagement with the telemedicine-based home monitoring system.

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Wellmann, MD, Phd student, Principal Investigator — Victor Babes Hospital for Infectious and Pulmonary Diseases, Timisoara, Romania
Locations (1):
- Dr. Victor Babeș Clinical Hospital for Infectious Diseases and Pulmonology, Timișoara, Timișoara, Timiș County, Romania

IPD SHARING:
Plan to Share IPD: No